CLINICAL TRIAL: NCT02151565
Title: High-tone External Muscle Stimulation for Treatment of Chronic Pain
Brief Title: High-tone External Muscle Stimulation for Pain Reduction
Acronym: HTEMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West German Center of Diabetes and Health (Other)
Collaborators: gbo Medizintechnik AG (Unknown)
Responsible Party: Principal Investigator, Stephan Martin, Principal investigator, West German Center of Diabetes and Health
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HTEMS
Record Dates: First submitted 2014-05-28; First posted 2014-05-30 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Chronic Radicular Back Pain; Lumboischialgia; Cervico Brachialgia
Keywords: back pain; sciatica; electrotherapy; HTEMS; TENS
MeSH Terms: conditions — Back Pain; Sciatica | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HTEMS (Experimental): High-tone external muscle stimulation 5 times within 10 days
  Interventions: Device: HTEMS
- TENS (Active Comparator): Transcutaneous electrical nerve stimulation 5 times within 10 days
  Interventions: Device: TENS

INTERVENTIONS:
Device: HTEMS
  Other Names: HITOP 191 (gbo Medizintechnik AG, Rimbach, Germany)
  Arms: HTEMS
Device: TENS
  Other Names: Dumo 2.4 (CEFAR Medical, Lund, Sweden)
  Arms: TENS

SUMMARY:
Sciatica is a common pain problem that affects not only the patient but also constitutes a socioeconomic burden and thus affects the whole society. So far, current pharmacologic therapies are inadequate for many patients. Therefore, we evaluated application of high-tone external muscle stimulation (HTEMS) compared to transcutaneous electrical nerve stimulation (TENS) on radicular pain associated with sciatica.

DETAILED DESCRIPTION:
Hospital patients (n=100) with chronic sciatica and stable oral analgesic regimen were included into this randomized controlled cross-over trial. Each intervention was administered for a period of 45 min 5 times within 10 days, with a 3-day wash-out period before cross-over. Health impairments had been assessed using the visual analog scales (VAS) for radicular pain before and after intervention and differences in radicular pain between groups were analysed with the Mann-Whitney test.

ELIGIBILITY:
Inclusion Criteria:

* sciatica due to degenerative spine disorders
* stable oral analgesic regimen

Exclusion Criteria:

* history of drug or alcohol abuse
* cardiac pacemaker or defibrillator
* pregnancy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Back pain | 10 days
  Back pain measured by an 11-point visual analogue scale (VAS) with 0 = none and 10 = worst pain imaginable

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - St. Vinzenz Krankenhaus, Düsseldorf
  - Düsseldorf Catholic Hospital Group, Düsseldorf